CLINICAL TRIAL: NCT00284102
Title: Positive End Expiratory Pressure (PEEP) Test and Gas Exchange in ALI/ARDS Patients
Brief Title: PEEP Test and Gas Exchange in ALI/ARDS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Davide Chiumello, Policlinico Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1700
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: gas exchange; dead space; respiratory failure; ALI/ARDS patients
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency | interventions — Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): ALI/ARDS patients
  Interventions: Procedure: Mechanical ventilation

INTERVENTIONS:
Procedure: Mechanical ventilation — measurement of gas exchange, dead space, respiratory mechanics 5, 15, 30, 60 minutes from PEEP change (5 and 15 cmH2O)

SUMMARY:
The investigators aim to study the effect of different levels of PEEP in ALI/ARDS patients on gas exchange.

DETAILED DESCRIPTION:
In a population of ALI/ARDS patients during mechanical ventilation we will evaluate the effect of different levels of PEEP on gas exchange and dead space.

ELIGIBILITY:
Inclusion Criteria:

* ALI/ARDS patients requiring mechanical ventilation

Exclusion Criteria:

* Hemodynamic instability
* Barotrauma

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Gas exchange, dead space, respiratory mechanics | 5, 15, 30, 60 minutes from PEEP change

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Principal Investigator — Policlinico Hospital
Locations (1):
- Policlinico Hospital, Milan, Italy